CLINICAL TRIAL: NCT04426669
Title: A Phase I/II Trial in Patients With Metastatic Gastrointestinal Epithelial Cancer Administering Tumor-Infiltrating Lymphocytes in Which the Gene Encoding CISH Was Inactivated Using the CRISPR/Cas9 System
Brief Title: A Study of Metastatic Gastrointestinal Cancers Treated With Tumor Infiltrating Lymphocytes in Which the Gene Encoding the Intracellular Immune Checkpoint CISH Is Inhibited Using CRISPR Genetic Engineering
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Intima Bioscience, Inc. (Industry)
Collaborators: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019LS002; NCT03538613 (obsolete NCT alias)
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Gastrointestinal Epithelial Cancer; Gastrointestinal Neoplasms; Cancer of Gastrointestinal Tract; Cancer, Gastrointestinal; Gastrointestinal Cancer; Colo-rectal Cancer; Pancreatic Cancer; Gall Bladder Cancer; Colon Cancer; Esophageal Cancer; Stomach Cancer
Keywords: Adoptive Cell Therapy, Immunotherapy, Gene Therapy, CISH checkpoint, CRISPR
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms; Gallbladder Neoplasms; Esophageal Neoplasms; Stomach Neoplasms | interventions — Cyclophosphamide; fludarabine; aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CISH CRISPR TIL / Phase I Arm (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine +escalating doses of CISH inactivated TIL + high-dose aldesleukin
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Tumor-Infiltrating Lymphocytes (TIL); Drug: Aldesleukin
- CISH CRISPR TIL / Phase II Arm (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + MTD of CISH inactivated TIL
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Tumor-Infiltrating Lymphocytes (TIL); Drug: Aldesleukin

INTERVENTIONS:
Drug: Cyclophosphamide — Day -6 and Day -5: Cyclophosphamide 60 mg/kg/dose as a 2 hour intravenous infusion with Mesna 15 mg/kg/dose, 1st dose prior to Cyclophosphamide infusion then at 3,6,9 and 12 hours later.
Drug: Fludarabine — Day -7 to Day -3 : Fludarabine 25 mg/m^2/dose as a 1 hour intravenous infusion per institutional guidelines once a day for 5 doses beginning on Day -7. Fludarabine will be started approximately 1 to 2 hours after the cyclophosphamide on Day -6 and Day -5.
Biological: Tumor-Infiltrating Lymphocytes (TIL) — Day 0 : Each bag of autologous CISH inactivated TIL for infusion will be administered intravenously (IV) on the Patient Care Unit over 10-20 minutes at assigned dose level.
Drug: Aldesleukin — Days 1-4 : Aldesleukin at 720,000 U/kg as an intravenous infusion, every 8 -12 hours but, no more than 24 hours apart as tolerated for up to 6 doses.
  Other Names: Interleukin-2, IL-2

SUMMARY:
A clinical trial to assess the safety and efficacy of genetically-engineered, neoantigen-specific Tumor Infiltrating Lymphocytes (TIL) in which the intracellular immune checkpoint CISH has been inhibited using CRISPR gene editing for the treatment of Gastro-Intestinal (GI) Cancer.

DETAILED DESCRIPTION:
Tumor Infiltrating Lymphocytes (TIL) have shown efficacy in certain cancers, principally in melanoma. Efficacy in more common solid tumors has been demonstrated via the selection of cancer neoantigen-specific TIL. Combination cell surface checkpoint inhibitor therapy has also been employed in an attempt to enhance the efficacy of these cell therapies. Genetic engineering of T cells to further increase anti-tumor activity is now possible.

CISH (Cytokine-induced SH2 protein) is a novel intra-cellular immune checkpoint and an important negative regulator of T-cell signaling and function. The inhibition of CISH in mouse anti-tumor lymphocytes results in a marked increase in the ability of these lymphocytes to mediate tumor regression following administration to tumor bearing mice.

Additionally, data in genetically-engineered, neoantigen-specific human T cells in which CISH was inhibited, showed enhanced TCR functional avidity and increased ability of these T cells to detect cancer specific mutations and mount robust polyfunctional cytokine immune responses against their cognate cancer antigens. Thus, these T cells appear to have a significant advantage in inducing anti-tumor responses compared to wild-type anti-tumor lymphocytes.

The researchers have developed and optimized a CRISPR/Cas9 based strategy for precise and efficient genetic engineering in primary human T-cells without sacrificing cell viability or function, allowing for inhibition of a heretofore undruggable intracellular checkpoint.

Thus, in this protocol, the researchers propose to inhibit the gene encoding the intracellular checkpoint target CISH in lymphocytes from patients with metastatic cancers that are selected for anti-tumor activity in order to evaluate the safety and efficacy of genetically engineered T cell therapy for solid tumors in the setting of novel checkpoint inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic gastrointestinal epithelial cancer with progressive disease following at least one first line standard therapy. When available, archived tissue from original diagnosis will be obtained for research related testing.
* Must have measurable disease per RECIST 1.1 with at least one lesion identified as resectable for TIL generation (minimum volume of tumor tissue required is 1 cm^2 as single mass or fragments) and at least one other lesion meeting the RECIST criteria for measurable to serve as an indicator of disease response. The location of the tumor for TIL generation and method used to obtain (i.e. laparoscopy, endoscopic ultra sound, etc.) will be determined based on an individual patient's disease.
* Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible. Patients must not be receiving systemic steroids.
* Brain metastases are assessed using the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria.
* Age ≥ 18 years and ≤ 70 years.
* Clinical performance status of ECOG 0 or 1.
* Serology testing within 3 months of study enrollment (tumor collection):

  * Seronegative for HIV antibody. (The investigational treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immunocompetence and thus may be less responsive to the study treatment and more susceptible to its toxicities.)
  * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
  * Seronegative for anti-HBc, HBV/HCV/HIV-1 NAT, anti-HTLV-I/II, anti-T.cruzi, West Nile Virus NAT, anti-CMV, and RPR. (Note: Other blood viral testing may be required as updated on the FDA website: https://www.fda.gov/BiologicsBloodVaccines/SafetyAvailability/TissueSafety/ucm095440.htm#approved)
* Hematology within 14 days of study enrollment:

  * Absolute neutrophil count > 1000/mm^3 without the support of filgrastim
  * WBC ≥ 3000/mm^3
  * Platelet count ≥ 75,000/mm^3
  * Hemoglobin > 8.0 g/dl. Subjects may be transfused to reach this cutoff.
* Adequate organ function within 14 days of study enrollment defined as:

  * Serum ALT and AST ≤ 5.0 x ULN
  * Serum creatinine ≤ 1.6 mg/dl
  * Total bilirubin ≤ to 2.0 mg/dl, except in patients with Gilbert's Syndrome, who must have a total bilirubin ≤ 3.0 mg/dl.
* More than four weeks must have elapsed since prior systemic therapy at the time the patient receives the preparative regimen, and acute toxicities must have recovered to Grade 1 or less (except for toxicities such as alopecia or vitiligo). Disease appropriate standard therapy is permitted between tumor collection and start of the fludarabine and cyclophosphamide. Investigational therapy is prohibited.

Note: Patients may have undergone minor surgical procedures within the 3 weeks of the start of preparative therapy as long as all toxicities have recovered to Grade 1 or less.

* Willing to undergo outpatient non-mobilized leukapheresis (3 hour collection) prior to the tumor collection
* Agrees to remain in the Twin Cities metropolitan area (within 1 hour drive of the University of Minnesota) after the CISH KO TILs infusion through the End of Treatment visit (Day 28)
* Voluntary written consent prior to the performance of any research related procedures

Exclusion Criteria:

* Pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant. Women of childbearing potential (defined as menses within previous 12 month and/or FSH ≤ 40 IU/L) must have a negative pregnancy test (serum or urine) within 7 days of enrollment. A repeat negative pregnancy test is required within 7 days of beginning the preparative chemotherapy.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Concurrent opportunistic infection (The treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune-competence may be less responsive to the treatment and more susceptible to its toxicities).
* Active systemic infections requiring anti-infective treatment, coagulation disorders or any other active major medical illnesses.
* Concurrent systemic steroid therapy.
* History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, or aldesleukin.
* History of coronary revascularization or ischemic symptoms.
* Documented LVEF ≤ 45% tested in patients:

  * Age ≥ 65 years and/or
  * With clinically significant atrial and/or ventricular arrhythmias, including but not limited to: atrial fibrillation, ventricular tachycardia, second- or third-degree heart block, or have a history of ischemic heart disease and/or chest pain. Patients < 65 years of age who present with cardiac risk factors (e.g., diabetes, hypertension, obesity) may undergo cardiac evaluation as noted above.
* Clinically significant patient history that in the judgment of the PI would compromise the patient's ability to tolerate high-dose aldesleukin.
* Documented FEV1 ≤ 50% predicted tested in patients with:

  * A prolonged history of cigarette smoking (approximately 20 packs/year within the past 2 years) and/or
  * Symptoms of respiratory dysfunction
* Receiving any investigational agents.

Confirmation of Eligibility Prior to CY/FU Start:

Due to a 10-12 week or more delay between study enrollment and the start of study treatment, the following eligibility criteria must be met:

* Clinical performance status of ECOG 0 or 1
* Hematology within 7 days of starting lymphodepleting chemotherapy:

  * Absolute neutrophil count > 1000/mm^3 without the support of filgrastim
  * WBC ≥ 3000/mm^3
  * Platelet count ≥ 100,000/mm^3
  * Hemoglobin > 8.0 g/dl. Subjects may be transfused to reach this cutoff.
* Adequate organ function within 7 days of starting lymphodepleting chemotherapy:

  * Serum ALT and AST ≤ 5.0 x ULN
  * Serum creatinine ≤ 1.6 mg/dl
  * Total bilirubin ≤ to 2.0 mg/dl, except in patients with Gilbert's Syndrome, who must have a total bilirubin ≤ 3.0 mg/dl.
* Seronegative for HIV antibody, hepatitis B antigen, and hepatitis C antibody as tested within 3 months of beginning lymphodepleting chemotherapy. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative
* More than four weeks must have elapsed since the last dose of prior systemic therapy and the start of the lymphodepleting chemotherapy, and acute toxicities must have recovered to Grade 1 or less (except for toxicities such as alopecia or vitiligo).
* Sexually active females of child-bearing potential and males with female partners of child-bearing potential must agree to use effective contraception for the duration of study treatment starting with the 1st dose of fludarabine and for 4 months after the last dose of aldesleukin. Examples of effective contraception includes an IUD or implant plus a condom. Women of non-childbearing potential are defined as those who have no uterus, ligation of the fallopian tubes, or permanent cessation of ovarian function due to ovarian failure or surgical removal of the ovaries. A woman also is presumed to be infertile due to natural causes if she has been amenorrheic for > 12 months and/or has an FSH > 40 IU/L.
* Negative pregnancy test within 7 days of starting lymphodepleting chemotherapy in women of childbearing potential.
* No change in medical status or social situation that would make study participation not in the best interest of the patient in the opinion of the enrolling investigator.
* Continues to agree to remain in the Twin Cities metropolitan area (within 1 hour drive of the University of Minnesota) after the CISH KO TILs infusion through the End of Treatment visit (Day 28)
* Voluntary signed the study treatment consent form within 28 days prior to the start of the lymphodepleting chemotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 28 Days Post IL-2
  Highest dose at which less than or equal to 1 of 6 patients experienced a DLT or the highest dose level studied if DLTs are not observed at any of the dose levels
Preliminary efficacy of tumor reactive autologous lymphocytes with knockout of CISH gene in patients with refractory metastatic gastrointestinal epithelial cancers: changes in diameter | Every 4 Weeks for the first three months, then every 8 weeks thereafter, up to 2 years
  Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST v1.1 criteria
Safety of tumor reactive autologous lymphocytes with knockout of the CISH gene - Incidence of Adverse Events | 2 Years or Disease Progression
  Incidence of Adverse Events

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 Years or Disease Progression
  Progression-Free Survival (PFS) of patients with metastatic gastrointestinal cancers treated using the autologous lymphocytes
Overall Survival (OS) | 2 Years or Disease Progression
  Overall Survival (OS) of patients with metastatic gastrointestinal cancers treated using the autologous lymphocytes
Toxicity profiles resulting from treatment using these engineered tumor-infiltrating lymphocytes | 2 Years or Disease Progression
  Incidence of targeted toxicities events

CONTACTS AND LOCATIONS:
Overall Officials: Emil Lou, MD, PhD, Principal Investigator — Division of Hematology, Oncology and Transplantation, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Palmer DC, Guittard GC, Franco Z, Crompton JG, Eil RL, Patel SJ, Ji Y, Van Panhuys N, Klebanoff CA, Sukumar M, Clever D, Chichura A, Roychoudhuri R, Varma R, Wang E, Gattinoni L, Marincola FM, Balagopalan L, Samelson LE, Restifo NP. Cish actively silences TCR signaling in CD8+ T cells to maintain tumor tolerance. J Exp Med. 2015 Nov 16;212(12):2095-113. doi: 10.1084/jem.20150304. Epub 2015 Nov 2. PMID 26527801
- [Background] Osborn MJ, Webber BR, Knipping F, Lonetree CL, Tennis N, DeFeo AP, McElroy AN, Starker CG, Lee C, Merkel S, Lund TC, Kelly-Spratt KS, Jensen MC, Voytas DF, von Kalle C, Schmidt M, Gabriel R, Hippen KL, Miller JS, Scharenberg AM, Tolar J, Blazar BR. Evaluation of TCR Gene Editing Achieved by TALENs, CRISPR/Cas9, and megaTAL Nucleases. Mol Ther. 2016 Mar;24(3):570-81. doi: 10.1038/mt.2015.197. Epub 2015 Oct 27. PMID 26502778
- [Background] Tran E, Ahmadzadeh M, Lu YC, Gros A, Turcotte S, Robbins PF, Gartner JJ, Zheng Z, Li YF, Ray S, Wunderlich JR, Somerville RP, Rosenberg SA. Immunogenicity of somatic mutations in human gastrointestinal cancers. Science. 2015 Dec 11;350(6266):1387-90. doi: 10.1126/science.aad1253. Epub 2015 Oct 29. PMID 26516200
- [Derived] Johnson MJ, Sumstad D, Folsom TD, Slipek NJ, DeFeo AP, Growe M, Kadidlo D, Thyagarajan B, Starr TK, Lou E, Choudhry M, Moriarity BS, Webber BR, McKenna DH. Clinical manufacture of CRISPR/Cas9-based cytokine-induced SH2 protein knock-out tumor-infiltrating lymphocytes for gastrointestinal cancers. Cytotherapy. 2025 Oct;27(10):1229-1239. doi: 10.1016/j.jcyt.2025.06.007. Epub 2025 Jun 21. PMID 40673842
- [Derived] Lou E, Choudhry MS, Starr TK, Folsom TD, Bell J, Rathmann B, DeFeo AP, Kim J, Slipek N, Jin Z, Sumstad D, Klebanoff CA, Ladner K, Sarkari A, McIvor RS, Murray TA, Miller JS, Rao M, Jensen E, Ankeny J, Khalifa MA, Chauhan A, Spilseth B, Dixit A, Provenzano PP, Pan W, Weber D, Byrne-Steele M, Henley T, McKenna DH, Johnson MJ, Webber BR, Moriarity BS. Targeting the intracellular immune checkpoint CISH with CRISPR-Cas9-edited T cells in patients with metastatic colorectal cancer: a first-in-human, single-centre, phase 1 trial. Lancet Oncol. 2025 May;26(5):559-570. doi: 10.1016/S1470-2045(25)00083-X. Epub 2025 Apr 29. PMID 40315882